CLINICAL TRIAL: NCT05166980
Title: Study of Multiply-fortified Salt Among Women of Reproductive Age and Preschool Children in India
Acronym: MFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); University of California, Davis (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MFS_1.2
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Nutrient Deficiency
Keywords: Micronutrient deficiencies
MeSH Terms: interventions — iodized salt; Iodine

STUDY DESIGN:
Intervention Model Description: 3-armed, double-blind, community-based efficacy trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study salts will be packaged in color-coded, polyethylene bags.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FePP-Q5S (Experimental): Salt fortified with iron in the form of ferric pyrophosphate (at 1.3 mg of iron per gram of salt) plus ethylenediaminetetraacetic acid (EDTA) as an enhancer of absorption, zinc in the form of zinc oxide (at 1.4 mg of zinc per gram of salt), vitamin B12 (at 0.6 ug of vitamin B12 per gram of salt), folic acid (at 52 ug per gram of salt) and iodine (at 30 mg of iodine per gram of salt). Mean intake of discretionary salt among women of reproductive age in the study area is 4.6 grams per day. Therefore, the FePP-Q5S will deliver an average of 6.0 mg of iron, 6.4 mg of zinc, 2.8 ug of vitamin B12, 241 ug of folic acid, and 138 mg of iodine to each participating woman per day.
  Interventions: Dietary Supplement: Mutiply-fortified salt
- eFF-Q5S (Experimental): Salt fortified with iron in the form of encapsulated ferrous fumarate (at 1.3 mg of iron per gram of salt), zinc in the form of zinc oxide (at 1.4 mg of zinc per gram of salt), vitamin B12 (at 0.6 ug of vitamin B12 per gram of salt), folic acid (at 52 ug per gram of salt) and iodine (at 30 mg of iodine per gram of salt). Mean intake of discretionary salt among women of reproductive age in the study area is 4.6 grams per day. Therefore, the eFF-Q5S will deliver an average of 6.0 mg of iron, 6.4 mg of zinc, 2.8 ug of vitamin B12, 241 ug of folic acid, and 138 mg of iodine to each participating woman per day.
  Interventions: Dietary Supplement: Mutiply-fortified salt
- Iodized Salt (Active Comparator): Iodized salt containing 30 mg of iodine per gram of salt. Mean intake of discretionary salt among women of reproductive age in the study area is 4.6 grams per day. Therefore, the iodized salt will deliver an average of 138 mg of iodine to each participating woman per day.
  Interventions: Dietary Supplement: Iodized salt

INTERVENTIONS:
Dietary Supplement: Mutiply-fortified salt — Salt fortified with iron, zinc, vitamin B12, folic acid, and iodine
  Other Names: Quintuply-fortified salt
  Arms: FePP-Q5S; eFF-Q5S
Dietary Supplement: Iodized salt — Salt fortified with iodine
  Other Names: Salt fortified with iodine
  Arms: Iodized Salt

SUMMARY:
Micronutrient (MN) deficiencies are highly prevalent in India, particularly among women of reproductive age (WRA) and preschool aged children (PSC). MN fortification of a staple food or condiment can be an effective strategy for improving the MN status of nutritionally vulnerable populations, as the approach is cost-effective, utilizes existing delivery systems, can deliver multiple MNs simultaneously, and does not require behavior change by the population. Salt is a particularly attractive vehicle for multiple MN fortification in India, as it is universally consumed in fairly consistent amounts; and 93% of households already use adequately iodized salt.

The overall goal of this study is to evaluate the nutritional impact of quintuply-fortified salt with iron in the form of FePP (FePP-Q5S, i.e. salt fortified with iron in the form of ferric pyrophosphate plus ethylenediaminetetraacetic acid as an enhancer of absorption; zinc in the form of zinc oxide; vitamin B12; folic acid; and iodine) vs. quintuply-fortified salt with iron in the form of eFF (eFF-Q5S i.e. salt fortified with iron in the form of encapsulated ferrous fumarate; zinc in the form of zinc oxide, vitamin B12, folic acid, and iodine) vs. iodized salt (IS) for the improvement of micronutrient status among nonpregnant WRA and preschool-aged children (12-59 months of age) in Punjab, India.

Enrolled women (and their affiliated households) will be randomized to receive 1 kg of their assigned study salt per month for 12 months, and will be instructed to use the study salt in place of their usual salt. Blood and urine samples will be collected from participant WRA and PSC at enrollment, 6 months and at the end of the 12-month intervention period. The change in the mean concentration of various MN biomarkers will be considered primary outcomes. Stool samples will also be collected from a subgroup of women and children to assess changes in the gut microbiome over the intervention period.

ELIGIBILITY:
Inclusion criteria for women of reproductive age:

1. 18-49 years of age;
2. Not currently pregnant (self-reported);
3. Not severely anemia (defined as a hemoglobin concentration < 8 g/dL);
4. Not planning to become pregnant within the next year;
5. Permanent resident of the study village with no plans to move or travel outside the village for more than 4 weeks over the next 12 months;
6. No serious health problems that requires regular visits to a health facility;
7. Willingness to use refined salt provided by the study as a primary source of household discretionary salt.

Exclusion criteria for women of reproductive age:

1. Age <18 or > 49 years of age;
2. Pregnant at the time of enrollment (self report) or planning to become pregnant within the next year;
3. Severely anemic (i.e. hemoglobin concentration < 8 g/dL);
4. Not a permanent resident of the study area;
5. Planning to leave the study area for at least one month over the study period;
6. Serious health problem that interferes with eating practices and/or requires hospitalization;
7. Unwilling to use refined salt provided by the study as the primary source of the household's discretionary salt.

Inclusion criteria for preschool children:

1. Child 12-59 months of age at the time of enrollment;
2. Child's mother or primary female caregiver has been enrolled into the parent trial;
3. Not severely anemic (defined as a hemoglobin concentration < 7 g/dL);
4. Child's family is a permanent resident of the study village with no plans to move or travel outside the village for more than 4 weeks over the next 12 months;
5. No serious medical problems that interfere with the child's eating practices;
6. Child's mother or primary female caregiver is willing to use refined salt provided by the study as the primary source of the household's discretionary salt for the course of the study.

Exclusion criteria for preschool children:

1. Child age < 12 or > 59 months of age;
2. Child's mother has not been enrolled in the parent trial;
3. Severely anemic (i.e. hemoglobin concentration < 7 g/dL);
4. Child's family is not a permanent resident of the study village and/or has plans to travel outside the village for more than 4 weeks over the next 12 months;
5. Serious health problem that interferes with the child's eating practices;
6. Child's mother or primary female caregiver is unwilling to use refined salt provided by the study as the primary sources of the household's discretionary salt for the course of the study.

Ages: 12 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1389 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Change in serum ferritin | Enrollment to 12 months (i.e. end of intervention period)
  Change in inflammation-adjusted mean serum ferritin concentration
Change in hemoglobin | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean hemoglobin concentration
Change in soluble transferrin | Enrollment to 12 months (i.e. end of intervention period)
  Change in inflammation-adjusted mean soluble transferrin concentration
Change in red blood cell folate | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean red blood cell folate concentration
Change in plasma zinc | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean plasma zinc concentration
Change in serum vitamin B12 | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean serum vitamin B12 concentration
Change in holo-transcobalamin | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean holo-transcobalamin concentration
Change in methylmalonic acid | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean concentration of methylmalonic acid
Change in serum folate | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean serum folate concentration
Change in urinary iodine | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean urinary iodine concentration
Change in serum thyroglobulin | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean serum thyroglobulin concentration

SECONDARY OUTCOMES:
Change in nail zinc | Enrollment to 12 months (i.e. end of intervention period)
  Change in mean fingernail zinc concentration
Change in gut microbiota | Enrollment to 12 months (i.e. end of intervention period)
  Change in the abundance of potentially beneficial microbiota in the gut

CONTACTS AND LOCATIONS:
Overall Officials: Christine McDonald, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
As soon as the manuscripts summarizing the study's primary outcomes are published, all datasets will be posted to Open Science Framework and made available to the public in accordance with the Gates Foundation's Open Data Policy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available as soon as the manuscripts summarizing the study's primary endpoints have been published. Data will be made available indefinitely.
URL: https://osf.io/

REFERENCES:
- [Derived] Thompson L, Goh YE, Jamwal M, Singh BL, Brar GK, Arnold CD, Westcott J, Long JM, Krebs NF, Zivkovic A, Das R, Duggal M, McDonald CM. The Effect of Quintuply-Fortified Salt on the Gut Microbiome of Young Children 1-5 y of Age in Punjab, India; A Substudy of a Randomized, Community-Based Trial. Curr Dev Nutr. 2025 Oct 23;9(11):107580. doi: 10.1016/j.cdnut.2025.107580. eCollection 2025 Nov. PMID 41323692
- [Derived] Goh YE, Duggal M, Das R, Manger MS, Jamwal M, Singh BL, Brar GK, Long JM, Westcott J, Thompson L, Arnold CD, Krebs NF, Brown KH, McDonald CM. Effects of quintuply-fortified salt on the micronutrient status of females of reproductive age in Punjab, India: a randomized, community-based trial. Am J Clin Nutr. 2025 Jul;122(1):146-156. doi: 10.1016/j.ajcnut.2025.04.009. Epub 2025 Jun 6. PMID 40610127
- [Derived] McDonald CM, Brown KH, Goh YE, Manger MS, Arnold CD, Krebs NF, Westcott J, Long JM, Gibson RS, Jamwal M, Singh BL, Dahiya N, Budhija D, Das R, Duggal M. Quintuply-fortified salt for the improvement of micronutrient status among women of reproductive age and preschool-aged children in Punjab, India: protocol for a randomized, controlled, community-based trial. BMC Nutr. 2022 Sep 6;8(1):98. doi: 10.1186/s40795-022-00583-y. PMID 36068647